CLINICAL TRIAL: NCT02197000
Title: A Nutritional Intervention to Decrease Breast Density Among Female BRCA Carriers -A Prospective Clinical Trial
Brief Title: A Nutritional Intervention to Decrease Breast Density Among Female BRCA (BReast CAncer Susceptibility Gene) Carriers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0117-14-RMC
Record Dates: First submitted 2014-07-20; First posted 2014-07-22 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2017-10

CONDITIONS: BRCA1 Gene Mutation; BRCA2 Gene Mutation
Keywords: BRCA mutation; Breast cancer; Estrogen metabolism; 3,3-Diindolylmethane; Breast density
MeSH Terms: conditions — Breast Neoplasms | interventions — 3,3'-diindolylmethane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DIM-Avail 100mg (Experimental): women will receive DIM 100mg*1/d, a nutritional supplement for 24 months.
  Interventions: Dietary Supplement: DIM-Avail 100mg

INTERVENTIONS:
Dietary Supplement: DIM-Avail 100mg — DIM 100 mg*1 daily for 2 years
  Other Names: 3,3-Diindolylmethane

SUMMARY:
The purpose of this study is to determine whether adding DIM supplement will decrease breast density among female BRCA mutation carriers in two years.

DETAILED DESCRIPTION:
The Research Question: In female BRCA mutation carriers, will adding DIM (100mg*1/d, a nutritional supplement), decrease breast density in two years?

Study design: A single center single arm prospective interventional study of the use of DIM to decrease risk of breast cancer among female BRCA carriers.

Study population: Subjects will be female carriers of a BRCA mutation and have more than 10% mammographic breast density at baseline.

Intervention: DIM supplement (100mg*1/d).

Study Time line: This will be a 2 years study. At initiation a breast mammography will be performed and eligibility assessed. Follow-up visits will occur every 4 months and quality of life questionnaires as well as adherence to DIM supplementation will be assessed. At the initiation and every 4 months blood and urine samples will be collected for Estrogen profile. At 12 and 24 months a mammography will be performed to verify changes in breast density.

Primary Endpoint: A decrease of more than 10% in breast density compared to baseline, following DIM supplementation intervention among female BRCA carriers.

Study impact: Decrease in mammographic breast density was shown to be a good marker for lower risk of breast cancer. This study has the potential to dramatically impact the management of female BRCA carriers. If we prove that by adding a food supplement breast density is decreased, we will change standard of care in these woman. In addition, the urine and blood samples collected during the study will be used for future translational research on the pathogenesis of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women who carrier the BRCA 1\2 mutation.
* No history of breast or ovarian malignancy.
* i. Baseline mammographic breast density is more than 10% OR ii. Baseline breast MRI with density or enhancement ≤ 2.
* Age 18-70.
* Absence of any psychological, familial, sociological or geographical situation potentially hampering adherence to the study protocol and follow-up schedule.
* Informed written consent must be signed according to ICH/EU GCP, before subject registration.

Exclusion Criteria:

* Women who have undergone preventive breast reduction.
* Breast imaging demonstrating a lesion suspected to be cancerous.
* Breast feeding or Pregnancy or planning to get pregnant.
* Known allergy to DIM and its ingredients.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-11-11 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Changes in breast density compared to baseline | 0, 12 and 24 months following intiation
  The amount of fibroglandular tissue (FGT) and background parenchymal enhancement (BPE) on magnetic resonance imaging (MRI)

SECONDARY OUTCOMES:
Estrogen profile | 0, 4, 8, 12, 16 and 24 months following initiation
  changes in TSH (Thyroid Stimulating Hormone), FSH (Follicle Stimulating Hormone), LH (Luteinizing Hormone), Estrogen, Prolactin, Progesterone and Testosterone compare to baseline
The Estronex Profile | 0, 12 and 24 months following initiation
  changes in the 2, 4, and 16 alpha- hydroxyderivative of estrone and the 2 and 4 methoxyestrone compare to baseline
change in Quality of life | 0, 4, 8, 12, 16 and 24 months following initiation
  Quality of life will be evaluate using the Revised Illness Perception Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: David Margel, MD, PhD, Principal Investigator — Rabin Medical Center, Beilinson campus, Petah-Tikva, Israel; Rinat Yerushalmi, MD, Principal Investigator — Rabin Medical Center, Beilinson Campus, Petah-Tikva, Israel
Locations (1):
- Rabin Medical Center, Beilinson Hospital, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No